CLINICAL TRIAL: NCT03231358
Title: Our Family Our Future: A Resilience-oriented Family Intervention to Prevent Adolescent HIV/STI Infection and Depression in South Africa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: University of Cape Town (Other); Desmond Tutu HIV Foundation (Other); Medical Research Council, South Africa (Other); Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Caroline Kuo, Assistant Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH114843 (NIH)
Record Dates: First submitted 2017-07-21; First posted 2017-07-27 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Human Immunodeficiency Virus; Depression; Sexually Transmitted Diseases
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Depression; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: We will randomize adolescents to an intervention arm (testing Our Family Our Future, n=440) or a control arm (n=440) of usual care (consisting of a packet of existing available brochures on HIV, STIs, mental health including places to access care). We will randomize based on permuted blocked randomization.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants randomized to the behavioral intervention called "Our Family Our Future." These participants will receive an intervention to prevent sexually transmitted infections (STIs) including HIV, Chlamydia trachomatis and Neisseria gonorrhoeae; sexual risk behavior; and depression onset. This is a behavioral intervention is delivered in a group setting over 3-4 consecutive weeks.
  Interventions: Behavioral: Our Family Our Future
- Control (No Intervention): The control arm will receive usual care (consisting of a packet of existing available brochures on HIV, STIs, mental health including places to access care).

INTERVENTIONS:
Behavioral: Our Family Our Future — Our Family Our Future is a 'selective' behavioral prevention program, designed to address HIV/STI acquisition, sexual risk behavior, and depression among adolescents (ages 14-16) in communities with high HIV prevalence and from families where adolescents and parents already exhibit mild, potentially troublesome, depressive symptoms but do not reach the threshold for further screening for a significant clinical depressive disorder. Participants receive the intervention in a community setting, in a facilitated group format. The intervention is comprised of 3-hour sessions, held weekly for 3 consecutive weeks with an individual family meeting in the third or fourth week depending on family desires.
  Arms: Intervention

SUMMARY:
The purpose of this study is to test the efficacy of Our Family Our Future, an integrated intervention for preventing HIV and depression onset among adolescents.

DETAILED DESCRIPTION:
Adolescent human immunodeficiency virus (HIV) and depression present significant public health challenges for South Africa, a country with the largest HIV epidemic globally and where structural factors including violence and poverty increase susceptibility for poor mental health. In families already experiencing psychological distress, adolescents face elevated risk for sexually transmitted infections (STIs) including HIV and depression. Preventive interventions are urgently needed during adolescence when risks for HIV, STIs, and depression in-crease exponentially. Preventive intervention strategies for adolescents should substantively involve families who can tailor prevention content to meet the unique needs of individual adolescents and reinforce formation and habituation of prevention behaviors. Moreover, evidence indicates common family risk and protective factors for adolescent HIV/STI risk behaviors and depression, underscoring the need for a family prevention approach. However, key gaps exist in family prevention science. In South Africa, few empirically supported family interventions integrate prevention of HIV/STI with depression for adolescents. This intervention (called Our Family Our Future) uses a resilience-oriented approach engages families in adolescent prevention from low-resource settings facing high adversity. The study will focus on adolescents (14-16 years) who are at an ideal developmental transition for family engagement in prevention. The age- and developmentally-tailored intervention - called Our Family Our Future - is based off of two empirically supported interventions that have been integrated and adapted to South Africa. In a pilot randomized trial, Our Family Our Future exhibited outstanding acceptability, feasibility and promising direction of effects including reductions of depressive symptoms; lower rates of sex; decreased unprotected sex; increased HIV testing; increased knowledge, motivation, intentions and self-efficacy for protective HIV/STI behaviors; improved family interactions; and increased resilience. Now investigators propose the next phase of this research program, an efficacy study of Our Family Our Future with three aims: (1) test the efficacy of the Our Family Our Future intervention in preventing HIV/STI acquisition among adolescents (14-16) with depressive symptoms by reducing HIV/STI risk behavior, and reducing depressive symptoms. The project will randomize N=880 adolescents to Our Family Our Future intervention or usual care with 6- and 12-month outcome assessments; (2) examine the extent to which the impact of the Our Family Our Future intervention is a) mediated by changes in resilience; behavioral skills; norms and attitudes relating to sex, condom use, gender; and family communication and functioning and b) moderated by the effect of sociodemographics, family HIV, and social protections; (3) identify barriers and facilitators to implementing Our Family Our Future within a large community-based organization setting with wide reach to provide data for future dissemination and scale-up.

ELIGIBILITY:
Inclusion Criteria:

* 14-16 years
* adolescent concurs that the adult identified is their parent (to also include primary caregivers in the pa-rental role)
* when more than one child in the family falls within the eligible age range, one child will be chosen at random
* lives in the household at least 4 days a week

Exclusion Criteria:

* no or low symptoms (<6) or clinically significant thresholds of depression (16+)

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1758 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Kuo, DPhil, MPhil, Principal Investigator — Brown University; Linda-Gail Bekker, MBChB, PhD, Principal Investigator — Desmond Tutu HIV Foundation; Dan J Stein, MBChB, PhD, Principal Investigator — University of Cape Town
Locations (1):
- Masiphumelele, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kuo C, Wasswa J, Orchowski L, Harrison A, Liu T, Sikweyiya Y, Berkowitz A, Adrian H, Rasmeni A, Mathews C. Rationale and design of a randomized controlled trial testing the efficacy of Safe South Africa, an intervention to prevent HIV risk behavior and sexual violence among adolescent boys. Trials. 2025 Dec 8;27(1):28. doi: 10.1186/s13063-025-09326-3. PMID 41361893

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention - Adolescents: Adolescents are the target participants for this study. Adolescent participants randomized to the behavioral intervention called "Our Family Our Future." These participants will receive an intervention to prevent sexually transmitted infections (STIs) including HIV, Chlamydia trachomatis and Neisseria gonorrhoeae; sexual risk behavior; and depression onset. This is a behavioral intervention, delivered in a group setting over 3-4 consecutive weeks.
  Our Family Our Future: Our Family Our Future is a 'selective' behavioral prevention program, designed to address HIV/STI acquisition, sexual risk behavior, and depression among adolescents (ages 14-16) in communities with high HIV prevalence and from families where adolescents and parents already exhibit mild, potentially troublesome, depressive symptoms but do not reach the threshold for further screening for a significant clinical depressive disorder. This intervention is delivered in a community setting, in a facilitated group format. The intervention is comprised of 3-hour sessions, held weekly for 3 consecutive weeks with an individual family meeting in the third or fourth week depending on family desires.
- Control - Adolescents: Adolescents are the target participants of this study. Adolescents assigned to the control arm will receive usual care (consisting of a packet of existing available brochures on HIV, STIs, mental health including places to access care).
- Intervention - Parents; Control - Parents: Adolescents are the target participants for this study. Parents are assigned into an arm, based on the assignment of their child). Because parents are not the primary target of the study, more minimal information is collected on them.
Period: Overall Study
Arm/Group | Intervention - Adolescents | Control - Adolescents | Intervention - Parents | Control - Parents
Started | 435 | 444 | 435 | 444
Completed | 391 | 434 | 389 | 432
Not Completed | 44 | 10 | 46 | 12

BASELINE CHARACTERISTICS:
Groups:
- Intervention - Adolescents: Participants randomized to the behavioral intervention called "Our Family Our Future." These participants will receive an intervention to prevent sexually transmitted infections (STIs) including HIV, Chlamydia trachomatis and Neisseria gonorrhoeae; sexual risk behavior; and depression onset. This is a behavioral intervention delivered in a group setting over 3-4 consecutive weeks.
- Control - Adolescents: The control arm will receive usual care (consisting of a packet of existing available brochures on HIV, STIs, mental health including places to access care).
- Total: Total of all reporting groups
Arm/Group | Intervention - Adolescents | Control - Adolescents | Intervention - Parents | Control - Parents | Total
Number analyzed (Participants) | 435 | 444 | 435 | 444 | 1758
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 435 | 444 | 435 | 444 | 1758
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Girl | 233 | 237 | 0 | 0 | 470
  Gender: Boy | 186 | 192 | 0 | 0 | 378
  Gender: Trans | 14 | 14 | 0 | 0 | 28
  Gender: Missing | 2 | 1 | 435 | 444 | 882
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black African | 404 | 409 | 404 | 409 | 1626
  Race: Coloured | 12 | 6 | 12 | 6 | 36
  Race: Indian or Asian | 1 | 3 | 1 | 3 | 8
  Race: White | 8 | 10 | 8 | 10 | 36
  Race: Other | 8 | 15 | 8 | 15 | 46
  Race: Missing | 2 | 1 | 2 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 435 | 444 | 435 | 444 | 1758
HIV Positive Status [Count of Participants; unit: Participants] — Population: The target of this intervention was adolescent participants. Thus, minimal information was collected on parent participants, to provide context for change (or lack of) in adolescent participants who are the target of the study/intervention.
  Participants
    number analyzed (Participants) | 435 | 444 | 0 | 0 | 879
    (all) | 0 | 2 |  |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of HIV and/or Chlamydia and/or Gonorrhoeae
Description: We will examine whether the intervention produces reductions in HIV and STI prevalence using biological tests for HIV, Chlamydia trachomatis, and Neisseria gonorrhoeae. We report on the prevalence of any HIV or STI (positive for one or more of HIV and/or Chlamydia and/or Neisseria).
Time Frame: 12 months
Population: We report on the prevalence of infection where the participant is at least positive for 1 HIV and/or STIs.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention: Participants randomized to the behavioral intervention called "Our Family Our Future." These participants will receive an intervention to prevent sexually transmitted infections (STIs) including HIV, Chlamydia trachomatis and Neisseria gonorrhoeae; sexual risk behavior; and depression onset. This is a behavioral intervention delivered in a group setting over 3-4 consecutive weeks.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 435 | 444
Participants | 60 | 70

2. Primary Outcome: Number of Participants Engaged In Vaginal Sex
Description: We will examine whether the intervention produces reductions in the number of participants engaged in vaginal sex and condom use.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 435 | 444
Participants
  Number of participants who had vaginal sex | 216 | 280
  Number of participants who used condoms in their last encounter of vaginal sex | 141 | 166

3. Primary Outcome: Depressive Symptoms
Description: We will examine whether the intervention produces reductions in depressive symptoms. Depressive symptoms will be measured through symptom scores on the Center for Epidemiologic Studies Depression Scale. Scores are summed, and range from 0 to 60. Higher scores correspond with worse depressive symptoms. There are ranges for the severity of depressive symptoms and these are as follows:
  0-15: May indicate no or low levels of depressive symptoms. 16 or higher: Suggests a risk for clinically significant depressive symptoms.
Time Frame: 12 months
Population: We captured symptom scores using the Center for Epidemiologic Studies Depression Scale. Scores are summed, and range from 0 to 60. Higher scores correspond with worse depressive symptoms. There are ranges for the severity of depressive symptoms and these are as follows:
  0-15: May indicate no or low levels of depressive symptoms. 16 or higher: Suggests a risk for clinically significant depressive symptoms.
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Intervention: Participants randomized to the behavioral intervention called "Our Family Our Future." These participants will receive an intervention to prevent sexually transmitted infections (STIs) including HIV, Chlamydia trachomatis and Neisseria gonorrhoeae; sexual risk behavior; and depression onset. This is a behavioral intervention involving adolescent-parent dyads, delivered in a group setting over 3-4 consecutive weeks.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 435 | 444
score on a scale | 18 [12 to 29] | 22 [12 to 29]

ADVERSE EVENTS:
Time Frame: We monitored any adverse events from enrollment of each participant, through study completion, approximately an average of 1 year in duration.
Description: The definition of adverse events and serious adverse events is consistent with out this is defined on clinicaltrials.gov
Groups:
- Intervention - Adolescents: Adolescents are the target participants for this study. Adolescent participants randomized to the behavioral intervention called "Our Family Our Future." These participants will receive an intervention to prevent sexually transmitted infections (STIs) including HIV, Chlamydia trachomatis and Neisseria gonorrhoeae; sexual risk behavior; and depression onset. This is a behavioral intervention, delivered in a group setting over 3-4 consecutive weeks.
Arm/Group | Intervention - Adolescents | Control - Adolescents | Intervention - Parents | Control - Parents
All-Cause Mortality (participants affected / at risk) | 0/435 | 0/444 | 0/435 | 0/444
Serious Adverse Events (participants affected / at risk) | 0/435 | 0/444 | 0/435 | 0/444
Other Adverse Events (participants affected / at risk) | 0/435 | 0/444 | 0/435 | 0/444

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT03231358/Prot_SAP_000.pdf